CLINICAL TRIAL: NCT03639987
Title: A Phase 2, Multicenter, Randomized, Parallel-Group, Double-Blind, Controlled Study of Aducanumab (BIIB037) in Subjects With Mild Cognitive Impairment Due to Alzheimer's Disease or With Mild Alzheimer's Disease Dementia to Evaluate the Safety of Continued Dosing in Subjects With Asymptomatic Amyloid-Related Imaging Abnormalities
Brief Title: A Study of Aducanumab in Participants With Mild Cognitive Impairment Due to Alzheimer's Disease or With Mild Alzheimer's Disease Dementia to Evaluate the Safety of Continued Dosing in Participants With Asymptomatic Amyloid-Related Imaging Abnormalities
Acronym: EVOLVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was discontinued based on futility analysis conducted on Phase 3 trials (NCT02477800 and NCT02484547) and not based on safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221AD205; 2018-002102-31 (EudraCT Number)
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Dysfunction; Alzheimer's Disease
Keywords: Aducanumab; BIIB037
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Aducanumab, intravenous infusion, every 4 weeks for up to Week 52 during the randomized treatment period. The dose will be titrated to a desirable dose. Participants will be managed for drug continuation and suspension. Following a 4-week follow-up period, eligible participants will continue to receive aducanumab, intravenous infusion, every 4 weeks for an additional 104 weeks in the long-term extension period.
  Interventions: Drug: Aducanumab; Drug: Placebo
- Group 2 (Experimental): Aducanumab, intravenous infusion, every 4 weeks for up to Week 52 during the randomized treatment period. The dose will be titrated to a desirable dose. Participants will be managed for drug continuation and suspension. Following a 4-week follow-up period, eligible participants will continue to receive aducanumab, intravenous infusion, every 4 weeks for an additional 104 weeks in the long-term extension period.
  Interventions: Drug: Aducanumab

INTERVENTIONS:
Drug: Aducanumab — Administered as specified in the treatment arm.
  Other Names: BIIB037
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Group 1

SUMMARY:
The primary objective of the study is to assess the safety impact of continuing aducanumab dosing in asymptomatic Amyloid-related Imaging Abnormalities (ARIA) in participants with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or with mild AD dementia. The secondary objective of the study is to characterize ARIA, from both the imaging and the clinical perspective and to characterize the safety, tolerability, pharmacokinetics (PK), and immunogenicity of aducanumab.

ELIGIBILITY:
Inclusion/ Exclusion Criteria

Key Inclusion Criteria:

* Ability of the participant or his/her legally authorized representative to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local participant privacy regulations.
* Must have at least 6 years of education or work experience to exclude mental deficits other than MCI due to AD or mild AD dementia.
* Must have evidence of cerebral Aβ accumulation, based on a positive PET scan of the brain. Previously obtained positron emission tomography (PET) scan (within 12 months of screening) is permissible. Previous PET scan images must be submitted to the central imaging vendor to confirm that study inclusion criteria are met.
* Must consent to apolipoprotein E (ApoE) genotyping.
* Must meet all of the following clinical criteria for MCI due to AD or mild AD dementia according to NIA-AA criteria [Albert 2011; McKhann 2011], and must have the following: MCI due to AD (a CDR global score of 0.5, and an MMSE score between 24 and 30 (inclusive)), or Mild AD dementia (a CDR global score of 0.5 or 1, and as MMSE score between 20 and 26 (inclusive)).

Key Exclusion Criteria:

* Any uncontrolled medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause of the participant's cognitive impairment (e.g., substance abuse, vitamin B12 deficiency, abnormal thyroid function, stroke or other cerebrovascular condition, Lewy body dementia, frontotemporal dementia, head trauma).
* Clinically significant unstable psychiatric illness (e.g., uncontrolled major depression, uncontrolled schizophrenia, uncontrolled bipolar affective disorder) within 6 months prior to Screening.
* Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening.
* Vaccinations within 10 days prior to randomization (Day 1).
* Female participants who are pregnant or currently breastfeeding.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (22):
- United States (22):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Pacific Research Network, Inc, San Diego, California
  - California Neuroscience Research Medical Group Inc., Sherman Oaks, California
  - JEM Research Institute, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Bioclinica Orlando, Orlando, Florida
  - Bioclinica Orlando, The Villages, Florida
  - Medical Research Health and Education Foundation, Inc, Columbus, Georgia
  - Josephson, Wallack, Munshower Neurology, P.C., Indianapolis, Indiana
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Advanced Memory Research Institute of NJ, PC, Toms River, New Jersey
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Neurology Clinic, PC, Cordova, Tennessee
  - Senior Adult Specialty Research, Austin, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
  - Kingfisher Cooperative, LLC, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 investigative sites in the United States from 20 December 2018 to 30 July 2019.
Pre-assignment Details: A total of 52 participants with Alzheimer's disease were enrolled in this study in one of the 2 groups: Group 1 and Group 2 to receive aducanumab titrated up to 10 mg/kg. The groups differed in the protocol specified management rules for amyloid-related imaging abnormalities (ARIA), in the event that moderate or severe asymptomatic ARIA was detected on MRI.
Groups:
- Group 1: Aducanumab dose titrated up to 10 mg/kg, IV infusion, following Group 1 ARIA management rules.
- Group 2: Aducanumab dose titrated up to 10 mg/kg, IV infusion, following Group 2 ARIA management rules.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 26 | 26
Completed | 0 | 0
Not Completed | 26 | 26
Not completed — Study terminated by sponsor | 26 | 25
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population is defined as all randomized participants who had received at least one dose of aducanumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.17) | 73.3 (7.14) | 72.9 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 26 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Impactful Amyloid-related Imaging Abnormalities (ARIA)
Time Frame: up to Week 54
Population: Clinically Impactful ARIA was to be assessed by an independent Adjudication Committee. At the time the study was terminated, the Adjudication Committee had not been formed; therefore, this outcome measure was not evaluated due to lack of data.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With ARIA by Severity as Obtained on Magnetic Resonance Imaging (MRI)
Description: ARIA by severity was obtained on Magnetic Resonance Imaging (MRI).
Time Frame: up to Week 54
Population: The safety population is defined as all randomized participants who had received at least one dose of aducanumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 26 | 26
Participants | 2 | 0

3. Secondary Outcome: Time to Onset of ARIA as Obtained on MRI
Time Frame: up to Week 54
Population: Due to small number of ARIA events, data is not reported due to participant confidentiality/human subjects protection assurances.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Resolution of ARIA as Obtained on MRI
Time Frame: up to Week 54
Population: as for outcome 3
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Symptomatic ARIA by Severity
Description: ARIA by severity was obtained on Magnetic Resonance Imaging (MRI).
Time Frame: up to Week 54
Population: The safety population is defined as all randomized participants who had received at least one dose of aducanumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 26 | 26
Participants | 1 | 0

6. Secondary Outcome: Time to Onset of Symptomatic ARIA
Time Frame: up to Week 54
Population: as for outcome 3
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Resolution of Symptomatic ARIA
Time Frame: up to Week 54
Population: as for outcome 3
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death, in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event), however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.
Time Frame: up to Week 54
Population: The safety population is defined as all randomized participants who had received at least one dose of aducanumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 26 | 26
Participants
  AEs | 15 | 9
  SAEs | 2 | 0

9. Secondary Outcome: Change From Baseline in the Montreal Cognitive Assessment (MoCA) at Week 54
Time Frame: Baseline, Week 54
Population: Due to early termination of the study, none of the participants reached the week 54 timepoint; therefore, data is not available for analysis.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Aducanumab Concentration in Serum
Time Frame: up to Week 54
Population: The safety population is defined as all randomized participants who had received at least one dose of aducanumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 26 | 26
Participants | 1 | 1

11. Secondary Outcome: Number of Participants With Antiaducanumab Antibodies in Serum
Time Frame: up to Week 54
Population: The safety population is defined as all randomized participants who received at least one dose of aducanumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 26 | 26
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 54
Description: The safety population is defined as all randomized participants who had received at least one dose of aducanumab.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/26
Other Adverse Events (participants affected / at risk) | 11/26 | 7/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=26) | Group 2 (N=26)
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=26) | Group 2 (N=26)
Headache (Nervous system disorders) | 5 | 4
Nasopharyngitis (Infections and infestations) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Study was discontinued based on futility analysis conducted on Phase 3 trials (NCT02477800 and NCT02484547). Enrolment and dosing was halted immediately upon the study termination announcement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03639987/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT03639987/SAP_001.pdf